CLINICAL TRIAL: NCT02505945
Title: The CALIBER Study Randomized Controlled Trial of LINX Versus Double-Dose Proton Pump Inhibitor Therapy for Reflux Disease
Acronym: CALIBER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Torax Medical Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 4959
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-12

CONDITIONS: GERD Gastroesophageal Reflux Disease
Keywords: Esophageal Reflux; Gastric Acid Reflux Disease; Heartburn
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (Active Comparator): Double-dose PPI [Omeprazole 20 mg BID (twice a day)]
  Interventions: Drug: Omeprazole
- Treatment Arm (Active Comparator): LINX Reflux Management System
  Interventions: Device: LINX Reflux Management System

INTERVENTIONS:
Drug: Omeprazole
  Other Names: Prilosec
  Arms: Control Arm
Device: LINX Reflux Management System
  Arms: Treatment Arm

SUMMARY:
This study compares mechanical sphincter augmentation (LINX Reflux Management System) to double-dose proton pump inhibitors (PPIs) for the management of reflux symptoms related to gastroesophageal reflux disease (GERD).

DETAILED DESCRIPTION:
Prospective, multicenter, 2:1 randomized, cross-over, two arms

* Control arm: Double-dose PPI [Omeprazole 20 mg BID (twice a day)]
* Treatment arm: LINX Reflux Management System Up to 20 study centers throughout the U.S. will participate. Approximately150 patients will be enrolled into the study. Subjects will be randomized 2:1 into the double-dose PPIs arm (100 subjects) and the LINX arm (50 subjects).

ELIGIBILITY:
Key Inclusion Criteria:

1. Patient seeks consultation for lack of satisfactory symptom response to once daily PPIs.
2. Age≥ 21 years old.
3. Abnormal distal esophageal pH determined by total % time pH <4 or DeMeester Score. Testing to be completed off GERD medications for at least 7 days, with the exception of antacids, which may be taken up until the morning of assessment.
4. Suitable surgical candidate (i.e. is able to undergo general anesthesia and laparoscopic surgery).
5. Patient has provided written informed consent for participation in the randomized study.

Key Exclusion Criteria:

1. Currently taking double-dose PPIs (twice daily dosing).
2. Hiatal hernia >3cm as determined by endoscopy.
3. Distal esophageal motility (average of sensors 3 and 4) is less than 35 mmHg peristaltic amplitude on wet swallows or <70% (propulsive) peristaltic sequences.
4. Esophagitis Grade C or D (Los Angeles classification).
5. Body mass index >35.
6. Diagnosed with an esophageal motility disorder LES.
7. Esophageal stricture or gross esophageal anatomic abnormalities
8. History of/or known Barrett's esophagus.
9. Suspected or known allergies to titanium, stainless steel, nickel or ferrous materials.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - University of South Alabama, Mobile, Alabama
  - Bapist Health, Heber Springs, Arkansas
  - University of Southern California, Los Angeles, California
  - UCSD, San Diego, California
  - SurgOne Foregut Institute, Englewood, Colorado
  - Albany Surgical PC, Albany, Georgia
  - Esophageal Institute of Atlanta, PC., Atlanta, Georgia
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Cuyuna Regional Medical Center, Crosby, Minnesota
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Adirondack Surgical Group, LLC, Saranac Lake, New York
  - University Hospitals Cleveland Medical Center - Geauga, Cleveland, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - The Oregon Clinic, Portland, Oregon
  - Albert Einstein Healthcare Network, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Scott and White Memorial Hospital, Round Rock, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Gundersen Lutheran, La Crosse, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rogers BD, Valdovinos LR, Crowell MD, Bell R, Vela MF, Gyawali CP. Number of reflux episodes on pH-impedance monitoring associates with improved symptom outcome and treatment satisfaction in gastro-oesophageal reflux disease (GERD) patients with regurgitation. Gut. 2021 Mar;70(3):450-455. doi: 10.1136/gutjnl-2020-321395. Epub 2020 May 28. PMID 32467089
- [Derived] Bell R, Lipham J, Louie BE, Williams V, Luketich J, Hill M, Richards W, Dunst C, Lister D, McDowell-Jacobs L, Reardon P, Woods K, Gould J, Buckley FP 3rd, Kothari S, Khaitan L, Smith CD, Park A, Smith C, Jacobsen G, Abbas G, Katz P. Magnetic Sphincter Augmentation Superior to Proton Pump Inhibitors for Regurgitation in a 1-Year Randomized Trial. Clin Gastroenterol Hepatol. 2020 Jul;18(8):1736-1743.e2. doi: 10.1016/j.cgh.2019.08.056. Epub 2019 Sep 10. PMID 31518717
- [Derived] Bell R, Lipham J, Louie B, Williams V, Luketich J, Hill M, Richards W, Dunst C, Lister D, McDowell-Jacobs L, Reardon P, Woods K, Gould J, Buckley FP 3rd, Kothari S, Khaitan L, Smith CD, Park A, Smith C, Jacobsen G, Abbas G, Katz P. Laparoscopic magnetic sphincter augmentation versus double-dose proton pump inhibitors for management of moderate-to-severe regurgitation in GERD: a randomized controlled trial. Gastrointest Endosc. 2019 Jan;89(1):14-22.e1. doi: 10.1016/j.gie.2018.07.007. Epub 2018 Jul 18. PMID 30031018

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 21 US clinical sites between July 2015 and February 2017
Period: Overall Study
Arm/Group | Control Arm | Treatment Arm
Started | 102 | 50
Completed | 80 | 46
Not Completed | 22 | 4
Not completed — Withdrawal by Subject | 13 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 2 | 1
Not completed — Lost to Follow-up | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Treatment Arm | Total
Number analyzed (Participants) | 102 | 50 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (13.7) | 47.8 (13.1) | 46.9 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 19 | 66
  Male | 55 | 31 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 1 | 8
  Not Hispanic or Latino | 95 | 49 | 144
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 93 | 48 | 141
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 102 | 50 | 152

OUTCOME MEASURES:

1. Primary Outcome: Elimination of Moderate-severe Regurgitation at 6 Months
Description: The primary endpoint was the percent of patients in both treatment arms who achieved elimination of moderate-severe regurgitation at 6 months, as reported on the foregut symptom questionnaire.
Time Frame: 6 months
Population: Excludes three subjects (2 LINX, 1 PPI) withdrawn following randomization and prior to either the implant procedure or start of double dose PPIs. One additional LINX subject in whom an implant was aborted due to device sizing issues was also excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 101 | 47
Participants | 10 | 42

2. Secondary Outcome: Percentage of Subjects With ≥50% Reduction in Total Gastroesophageal Reflux Disease-Health Related Quality of Life (GERD-HRQL) Scores
Description: Successful Reduction at 6 months (≥50% reduction in total) Gastroesophageal Reflux Disease-Health Related Quality of Life (GERD-HRQL) scores from Baseline PPI On medication GERD HRQL scores.
Time Frame: 6 months
Population: All available follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 87 | 47
Participants | 7 | 38

ADVERSE EVENTS:
Time Frame: 6 months
Description: For the purposes of this study, a reportable event will be defined as any untoward medical occurrence which has a strong relationship to the LINX device and/or implant procedure or PPI and another etiology is unlikely.
Arm/Group | Control Arm | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/102 | 1/50
Other Adverse Events (participants affected / at risk) | 10/102 | 24/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=102) | Treatment Arm (N=50)
Esophageal spasms (Gastrointestinal disorders) | 0 (0) | 1 (1) — resolved
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=102) | Treatment Arm (N=50)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 15 (16)
Bloating/gas (Gastrointestinal disorders) | 1 (2) | 4 (5)
Nausea (General disorders) | 3 (3) | 4 (4)
Chest pain (General disorders) | 0 (0) | 4 (4)
Esophageal spasms (Gastrointestinal disorders) | 0 (0) | 4 (4)
Epigastric pain or pressure (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal Pain (General disorders) | 3 (4) | 1 (1)
Implant site pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Belching (General disorders) | 1 (1) | 2 (2)
Odynophagia (General disorders) | 0 (0) | 1 (1)
Soreness (General disorders) | 1 (1) | 1 (1)
Diarrhea (General disorders) | 1 (1) | 1 (1)
Medication reaction (General disorders) | 2 (2) | 0 (0)
Worsening reflux (General disorders) | 2 (2) | 0 (0)
Arrythemia (Cardiac disorders) | 0 (0) | 1 (1)
Bone ache (General disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Change in voice (General disorders) | 0 (0) | 1 (1)
Constipation (General disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1)
Hiccups (General disorders) | 0 (0) | 1 (1)
Hoarseness (General disorders) | 0 (0) | 1 (1)
Inability to belch (General disorders) | 0 (0) | 1 (1)
Inability to vomit (General disorders) | 0 (0) | 1 (1)
Abnormal Manometric Outflow (General disorders) | 0 (0) | 1 (1)
Regurgitation (General disorders) | 1 (1) | 0 (0)
Vomiting (General disorders) | 0 (0) | 1 (1)
Worsening esophagitis (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must provide sponsor copy of any proposed publication at least (45)days prior to the submission. PI shall defer any publication until release of the publication of the results of the Study by the sponsors joint publication committee. In the event that a multiple center publication is not submitted within 12 mo. after the completion at all centers, PI may publish Study results from their individual experience, after submitting to Sponsor for review (90)days prior to submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT02505945/Prot_SAP_000.pdf